CLINICAL TRIAL: NCT04179669
Title: A Study to Evaluate Safety and Efficacy of IBI306 in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Safety and Efficacy of IBI306 in HeFH Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI306C301
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Heterozygous Familial Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI306 (Experimental): Participants received IBI306 150 mg subcutaneously Q2W or 450mg Q4W for 12 weeks.
  Interventions: Drug: IBI306
- placebo (Experimental): Participants received Placebo 150 mg subcutaneously Q2W or 450mg Q4W for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IBI306 — Administered by subcutaneous injection
  Arms: IBI306
Drug: placebo — Administered by subcutaneous injection
  Arms: placebo

SUMMARY:
IBI306 is a fully human monoclonal antibody that binds proprotein convertase substilisin/kexin type 9 (PCSK-9), preventing its interaction with the low-density lipoprotein cholesterol receptor (LDL-R) and thereby restoring LDL-R recycling and low-density lipoprotein cholesterol (LDL-C) uptake. In the phase I study, IBI306 was shown to be safe and well tolerated. There was robust reduction in LDL-C, Apo(B), non-HDL-C and lipoprotein (a) in healthy subjects. This study is a randomized, double-blind, placebo-controlled, repeated-dosing, multiple ascending dose trial to evaluate the efficacy and safety of a novel PCSK-9 anti-body, IBI306, in Chinese patients with heterozygous familial hypercholesterolemia.

DETAILED DESCRIPTION:
The study plans to enroll 148 patients with heterozygous familial hypercholesterolemia. Subjects will maintain a low-fat diet and stable current lipid-lowering therapy for at least 4 weeks and will be randomized into different dose groups at a 1:1 ratio, followed by a 2:1 randomization double-blind treatment with subcutaneous IBI306 150 mg (n=49) or placebo (n=25) every two weeks; or subcutaneous injection of IBI306 450mg (n=49) or placebo (n=25) every four weeks. Treatment lasts for 12 weeks. After 12 weeks, each group enters a 12-week open-label treatment, in which IBI306 subjects continue to receive IBI306, and placebo subjects shift to receive IBI306. The primary endpoint is the percent change in LDL-C levels relative to baseline at 12 weeks. Secondary endpoints include changes in baseline lipid levels, drug safety, and immunogenicity at 12 weeks and 24 weeks. The exploratory endpoint is the population pharmacokinetic profile of IBI306 in Chinese subjects with heterozygous familial hypercholesterolemia. If necessary, the dose of IBI306 will be adjusted accordingly based on the results of the ongoing multi-dose escalation study. After the open period, the subjects will be given a safety visit for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

• Subjects must meet all of the following inclusion criteria in order to be included in the study:

* Provide a signed and dated informed consent form
* Men or women 18 to 70 years of age at screening
* Weight ≥ 40 kg during screening
* Confirmed diagnosis of heterozygous familial hypercholesterolemia
* Maintain a low-fat diet and stabilize the current lipid-lowering therapy

Exclusion Criteria:

• Subjects who do not meet any of the following exclusion criteria cannot be included in the study:

* Patients diagnosed as homozygous familial hypercholesterolemia
* Dialysis or plasmapheresis performed within 4 months prior to screening
* History of liver transplant
* Subjects adjusted for treatment of statins, ezetimibe, niacin, omega-fatty acids within 4 weeks prior to screening
* New York Heart Association (NYHA) grade III or IV heart failure, or recent detection of left ventricular ejection fraction ≤ 30%
* Have serious cardiovascular, cerebrovascular, liver and kidney related diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of LDL-C decreased from baseline injection. | at 12 weeks

SECONDARY OUTCOMES:
Percentage change of LDL-C from baseline | to 24 weeks
Changes in LDL-C levels relative to baselin | at 12 and 24 weeks
The proportion of patients with LDL-C that were 50% lower than baseline | by 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Chai M, He Y, Zhao W, Han X, Zhao G, Ma X, Qiao P, Shi D, Liu Y, Han W, An P, Li H, Yan S, Ma Q, Deng H, Qian L, Zhou Y; CREDIT-2 investigators. Efficacy and safety of tafolecimab in Chinese patients with heterozygous familial hypercholesterolemia: a randomized, double-blind, placebo-controlled phase 3 trial (CREDIT-2). BMC Med. 2023 Feb 28;21(1):77. doi: 10.1186/s12916-023-02797-8. PMID 36855099